CLINICAL TRIAL: NCT05178914
Title: Personalized Medicine Using Coronary Microvascular Function Measured in Patient With Percutaneous Coronary Intervention in Angina
Acronym: DECISIONING
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 38RC21.0339
Record Dates: First submitted 2021-10-20; First posted 2022-01-05 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Coronary Microvascular Disease
Keywords: index of microcirculatory resistance
MeSH Terms: conditions — Microvascular Angina

STUDY DESIGN:
Intervention Model Description: Patients with a symptomatology of angina pectoris who have at least one epicardial lesion greater than or equal to 50% on coronary angiography evaluation
  The interventional group is defined by the disclosure of the IMR value. The initial IMR is used to guide therapy.
  The control group is defined as follows: the initial IMR has been performed but its result is not undisclosed (sham procedure) ; patients will receive standard medical treatment according to the physician's preference.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The interventional group (Experimental): Patients are defined by the disclosure of the IMR value. The initial IMR is used to guide therapy.
  For patients with initial IMR ≥ 25 will benefit from intensified coronary artery disease treatment to manage the microcirculatory damage according to the recommendations and consensus of European experts.
  For patients with a initial IMR < 25 will benefit from de-escalade therapeutic adaptation.
  Interventions: Procedure: Treatment adaptation
- The control group (Sham Comparator): The control group is defined as follows: the initial IMR has been performed but its result is not undisclosed (sham procedure) ; patients will receive standard medical treatment according to the physician's preference.
  Interventions: Procedure: Treatment adaptation

INTERVENTIONS:
Procedure: Treatment adaptation — Patients will benefit from intensified treatment or de escalation treatment according to the result of the index of microcirculatory resistance

SUMMARY:
The evidence demonstrating the importance of coronary microcirculation in the management of patients with coronary artery disease is growing. For example, in recent years, a number of studies have demonstrated that the presence of coronary microvascular disease (CMVD) contributes to increased cardiovascular morbidity and mortality independent of the extent and severity of coronary epicardial disease. The index of microcirculatory resistance (IMR) is an invasive index proposed for the diagnosis of CMVD. The ability of IMR to motivate therapeutic changes in order to subsequently reduce symptoms and improves the quality of life of our patients with stable coronary artery disease (CAD) was recently demonstrated. The prognostic value of IMR has also been shown in stable CAD with PCI. Thus, after optimal epicardial evaluation and if necessary revascularization according to FFR, IMR could represent a tool for personalized medicine adapted to the presence of severe CMVD.

The aim of the study is to demonstrate a positive effect of personalized medicine on angina in patients with epicardial coronary network lesion assessment by FFR and with significant CMVD assessed by IMR.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years
* Symptomatology of angina pectoris
* Receiving invasive coronary angiography
* FFR and microcirculatory resistance index (MRI) measurement for at least one epicardial lesion ≥ 50% :
* For lesions with FFR ≤ 0.8, revascularization with the XIENCE Sierra stent and its evolutions will be performed. Optimization of this epicardial revascularization will be evidenced by a post-PCI FFR > 0.8 on all major trunks and if an FFR measurement is not performed, absence of 50% or greater stenosis on two orthogonal views by quantitative coronary angiography [QCA] at the revascularization site.
* For lesions with FFR > 0.8 revascularization will not be performed
* Written informed consent

Exclusion Criteria:

* A non-coronary indication for coronary angiography, e.g. valve disease, hypertrophic obstructive cardiomyopathy.
* Severe renal dysfunction (GFR < 30 ml/min)
* Contraindications for adenosine: asthma, Second or third degree AV block without pacemaker or sick sinus syndrome, Systolic blood pressure less than 90 mm Hg, Recent use of dipyridamole or drugs containing dipyridamole, Methyl xanthenes such as caffeine aminophylline or theobromine block the effect of adenosine and should be stored at least 12 hours before testing, Known hypersensitivity to adenosine.
* Pregnant women, parturients and breastfeeding mothers
* Persons of full age who are subject to a legal protection measure or who are unable to express their consent
* Patient in a period of exclusion from another study
* Patient under administrative or judicial supervision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2022-03-31 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
The mean difference in angina severity | One year
  Assessed by the Seattle Angina Questionnaire summary score) between patients with an IMR ≥ 25 in the interventional group, benefiting from personalized medicine, and patients with IMR ≥ 25 in the control group benefiting from standard care

SECONDARY OUTCOMES:
To demonstrate a positive effect of personalized medicine guided by IMR assessment on physical limitation due to angina | At 6 months and 1 year
  The physical limitation scale is assessed by question 1 of the Seattle Angina questionnaire and measures how daily activities are limited by symptoms of coronary disease.
  This question includes 9 sub-questions with 5 possible answers from the worse to the best.
  The analysis will be performed between :
  * IMR ≥ 25 in the interventional group versus patients with an IMR ≥ 25 in the control group
  * IMR < 25 in the interventional group versus patients with an IMR < 25 in the control group
To demonstrate a positive effect of personalized medicine guided by IMR assessment on stability of angina | At 6 months and 1 year
  The angina stability scale is assessed by question 2 of the Seattle Angina Questionnaire and measures change in the frequency of angina at patient's most streneous level of activity.
  There are 5 possible answers from the worse to the best.
  The analysis will be performed between :
  * IMR ≥ 25 in the interventional group versus patients with an IMR ≥ 25 in the control group
  * IMR < 25 in the interventional group versus patients with an IMR < 25 in the control group
To demonstrate a positive effect of personalized medicine guided by IMR assessment on frequency of angina | At 6 months and 1 year
  The angina frequency scale is assessed by question 3 and 4 of the Seattle Angina questionaire. It measures the frequency of angina (question 3) and the need of nitroglycerin (question 4) For each question, there are 5 possible answers from the worse to the best.
  The analysis will be performed between :
  * IMR ≥ 25 in the interventional group versus patients with an IMR ≥ 25 in the control group
  * IMR < 25 in the interventional group versus patients with an IMR < 25 in the control group
To demonstrate a positive effect of personalized medicine guided by IMR assessment on perception of the disease. | At 6 months and 1 year
  Perception of illness will be analyzed by questions 9-11 of the Seattle Angina questionnaire and characterizes the illness-related burden experienced by the patient.
  The analysis will be performed between :
  * IMR ≥ 25 in the interventional group versus patients with an IMR ≥ 25 in the control group
  * IMR < 25 in the interventional group versus patients with an IMR < 25 in the control group
To demonstrate a positive effect of personalized medicine guided by IMR assessment with satisfaction with the treatment. | At 6 months and 1 year
  Satisfaction with the treatment is assessed by questions 5 to 8 of the Seattle Angina Questionnaire and quantifies patient's satisfaction with their current treatment.
  The analysis will be performed between :
  * IMR ≥ 25 in the interventional group versus patients with an IMR ≥ 25 in the control group
  * IMR < 25 in the interventional group versus patients with an IMR < 25 in the control group
To demonstrate a positive effect of personalized medicine guided by IMR on assessment of dyspnea. | At 6 months and 1 year
  The assessment of dyspnea will be evaluated by the Rose Dyspnea Scale, a 4-part questionnaire.
  The analysis will be performed between :
  * IMR ≥ 25 in the interventional group versus patients with an IMR ≥ 25 in the control group
  * IMR < 25 in the interventional group versus patients with an IMR < 25 in the control group
To demonstrate a positive effect of personalized medicine guided by IMR assessment on quality of life. | At 6 months and 1 year
  The assessment on quality of life will be evaluated by the EQ5D-5L, a 5-part questionnaire.
  The analysis will be performed between :
  * IMR ≥ 25 in the interventional group versus patients with an IMR ≥ 25 in the control group
  * IMR < 25 in the interventional group versus patients with an IMR < 25 in the control group
To demonstrate a positive effect of personalized medicine guided by IMR assessment on health care consumption. | 1 year
  Health care consumption will be assessed by the number and relative cost of consultations with a general practitioner, cardiologist or other specialist; as well as the number of imaging tests performed. These examinations will be collected by self-reporting at the time of follow-up visits.
  The analysis will be performed between :
  * IMR ≥ 25 in the interventional group versus patients with an IMR ≥ 25 in the control group
  * IMR < 25 in the interventional group versus patients with an IMR < 25 in the control group
To demonstrate a positive effect of personalized medicine guided by IMR assessment on the number of Major Cardiovascular Events (MACE). | 1 year
  MACE will be assessed by cumulative rates in the year of death, myocardial infarction, target vessel failure, hospitalization for unstable angina, or heart failure.
  The analysis will be performed between :
  * IMR ≥ 25 in the interventional group versus patients with an IMR ≥ 25 in the control group
  * IMR < 25 in the interventional group versus patients with an IMR < 25 in the control group
To demonstrate a positive effect of personalized medicine guided by IMR assessment on the prevalence of subgroups. | At 6 months and 1 year
  The prevalence of sub-groups will be assessed by performing IMR pre and post-PCI for each patient.
To demonstrate a positive effect of personalized medicine guided by IMR assessment on the angina Severity according to subgroups. | At 6 months and 1 year
  The angina Severity will be assessed by The Seattle Angina Questionnaire.
  The analysis will therefore be performed between subgroups as follow:
  * IMR pre-PCI <25 and IMR post-PCI <25
  * IMR pre-PCI <25 and IMR post-PCI ≥25
  * IMR pre-PCI ≥25 and IMR post-PCI <25
  * IMR pre-PCI ≥25 and IMR post-PCI ≥25

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Grenoble Alpes, La Tronche, France

IPD SHARING:
Plan to Share IPD: No